CLINICAL TRIAL: NCT06944522
Title: exPDite-2: A Phase 3 Study to Assess the Efficacy and Safety of Midbrain Dopaminergic Neuronal Cell Therapy (Bemdaneprocel) for Participants With Parkinson's Disease
Brief Title: A Study to Investigate the Efficacy and Safety of Bemdaneprocel in Adults Who Have Parkinson's Disease
Acronym: exPDite-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BlueRock Therapeutics (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRT-DA01-301
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Parkinsons Disease (PD)
Keywords: exPDite-2; Cell Therapy; Cellular Therapy; Dopaminergic Neuronal Cell Therapy; Parkinsons Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In the double-blind period, participants will be randomized at a 2:1 ratio to either receive bemdaneprocel or undergo sham surgery. Participants will receive immunosuppression or placebo equivalents for approximately 12 months. Approximately 18 months after the last participant is enrolled and based on the results of the primary analysis and review by the independent data monitoring committee (DMC), eligible participants who underwent sham surgery and remain actively enrolled in the study will have the opportunity to receive bemdaneprocel in the open-label period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Bemdaneprocel will be administered on Day 0
  Interventions: Biological: bemdaneprocel
- Group B (Sham Comparator): Sham surgery will be performed on Day 0
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Biological: bemdaneprocel — Investigational cell therapy comprising midbrain dopaminergic neuron progenitors derived from human embryonic stem cells
  Other Names: MSK-DA01; BRT-DA01
  Arms: Group A
Procedure: Sham surgery — Sham surgery will be performed on Day 0
  Arms: Group B

SUMMARY:
Study BRT-DA01-301 is a Phase 3 multicenter, randomized, sham surgery-controlled, double-blind study to assess efficacy and safety of bemdaneprocel in approximately 102 adults with Parkinson's Disease (PD).

DETAILED DESCRIPTION:
The BRT-DA01-301 study is a Phase 3, multicenter, randomized, sham surgery-controlled, double-blind study involving approximately 102 participants with Parkinson's Disease (PD). Participants will be randomized in a 2:1 ratio to either receive bemdaneprocel or undergo sham surgery. The study includes an immunosuppression regimen and placebo equivalents to maintain blinding. The primary objective is to evaluate the efficacy of bemdaneprocel on motor symptoms in participants with PD. The secondary objective is to evaluate the effects of bemdaneprocel on Motor function, Quality of life, Non-motor symptoms of PD, Disease severity, and Use of PD medications or therapies compared with participants who undergo sham surgery. Participants will be followed for at least 18 months in the double-blind period and up to five years if they receive bemdaneprocel.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically established PD as defined by the International Parkinson and Movement Disorders Society
* Individual of any sex ≥45 to ≤75 years of age at informed consent
* Robust and clear response to DA therapy as defined by MDS-UPDRS Part III
* ≥4 and <12 years from time of PD diagnosis at informed consent
* Must demonstrate responsiveness to levodopa therapy
* Receiving medical therapy for the treatment of PD symptoms
* ≥2.5 hours of daily OFF-time
* Vaccinated per current national guidelines or local practice for patients with altered immunocompetence

Exclusion Criteria:

* PD presenting with recurrent falls
* Diagnosis of primary mitochondrial disorder, epilepsy, stroke, multiple sclerosis, or clinical features suggestive of a neurodegenerative disease other than PD, including multiple system atrophy, progressive supranuclear palsy, corticobasal degeneration, or Lewy body dementia
* Any current or relevant previous history of serious, severe, or unstable physical, neurological, or psychiatric illness that may interfere with study participation, participant's safety, or assessment of endpoints per investigator's judgment
* History of gene therapy or cell therapy
* Prior treatment with intrajejunal or subcutaneous infusion therapies for PD
* Prior surgical or radiation therapy to the brain, including deep brain stimulation (DBS) and lesion therapy, or prior history of intradural spinal cord surgery
* Contraindication to surgery, general anesthesia, cell therapy, immunosuppression, or other required drugs, or anything that prevents use of PET or MRI
* Any active infection (including but not limited to HIV, HCV, HBV, CMV, syphilis, or tuberculosis) or condition that, in the opinion of the investigator could put the participant at significant risk from immunosuppression or impact the participant's ability to perform study assessments
* Current or previously active malignant disease within the past 5 years
* Chronic immunosuppressive therapy
* Receipt of another investigational therapy within 5 half-lives of the active treatment
* Pregnancy or breastfeeding

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in PD diary measure of ON-time without troublesome dyskinesia, adjusted for a 16-hour waking day | From baseline to Week 78

SECONDARY OUTCOMES:
Change from baseline in PD diary measure of OFF-time, adjusted for a 16-hour waking day | From baseline to Week 78
Change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score in the off-medication state. Part III score can range from 0 to 132, with lower scores being better. | From baseline to Week 78
Change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II score. Part II score can range from 0 to 52, with lower scores being better. | From baseline to Week 78
Change from baseline in Parkinson's Disease Questionnaire-39 (PDQ-39) summary index. Summary index score can range from 0 to 100, with lower scores being better. | From baseline to Week 78
Incidence and severity of treatment-emergent adverse events | From baseline to month 60

CONTACTS AND LOCATIONS:
Locations (29):
- United States (22):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA NeuroTranslational Research Center, Los Angeles, California
  - University of Colorado Hospital - Neurology Clinic, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Health System - Neurology, Miami, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Parkinson's Disease and Movement Disorders Center at Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Tufts Medical Center - Neurology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Clinical Research Unit - Neurology, Ann Arbor, Michigan
  - University of Michigan Clinical Research Unit - Neurology, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - UBMD Neurology, Buffalo, New York
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - Rhode Island Hospital - Neurology, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - EvergreenHealth - Research Department, Kirkland, Washington
- Australia (6):
  - NeuRA (Neuroscience Research Australia), Randwick, New South Wales
  - Gold Coast Hospital & Health Service, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- CHUM - Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada